CLINICAL TRIAL: NCT05935215
Title: A Multicenter, Single Arm, Open-label Study to Evaluate Efficacy and Safety of Switching From Anti-C5 Antibody Treatment to Iptacopan Treatment in Study Participants With aHUS
Brief Title: Efficacy and Safety of Switching From Anti-C5 Antibody Treatment to Iptacopan Treatment in Study Participants With Atypical Hemolytic Uremic Syndrome (aHUS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023F12302
Expanded Access: NCT05222412 (Available)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: Atypical Hemolytic Uremic Syndrome; aHUS, thrombotic microangiopathy; TMA
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Thrombotic Microangiopathies | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iptacopan 200 mg b.i.d. (Experimental): open label arm of iptacopan 200 mg b.i.d.
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Open Label
  Other Names: LNP023

SUMMARY:
The purpose of this Phase 3 study is to evaluate the efficacy and safety of iptacopan upon switching from anti-C5 antibody to iptacopan treatment in study participants with aHUS.

DETAILED DESCRIPTION:
The study is designed as a multicenter, single-arm, open label study to evaluate the efficacy and safety of iptacopan upon switching from anti-C5 antibody to iptacopan treatment in participants with aHUS. It consists of a screening period of up to 8 weeks followed by a 12-Month Core Treatment period and 12-Month Extension Treatment period.

The study will assess the effects of iptacopan on a range of efficacy assessments relevant to aHUS.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult participants ≥ 18 years of age with diagnosis of aHUS for whom etiologies of other types of TMA and non-aHUS kidney disease have been excluded.
* Currently on the recommended weight-based dosage regimen of anti-C5 antibody treatment for at least 3 months prior to the screening visit.
* Clinical evidence of response to anti-C5 antibody treatment (in absence of PE/PI) for at least 3 months prior to entering the screening period as defined by:

  1. Hematological normalization in platelet count ≥150 x 109/L and LDH below upper limit of normal [ULN], and
  2. Stable or improving kidney function as defined by ≤15% increase in serum creatinine.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infections is required prior to the start of treatment with iptacopan.
* If not received previously or if a booster is required, vaccination against Haemophilus influenzae infection, should be given, if available and according to local regulations.

Exclusion Criteria:

* History of aHUS disease relapse while on anti-C5 antibody treatment.
* eGFR < 30 ml/min/1.73m^2
* Active infection or history of recurrent invasive infections caused by encapsulated bacteria, i.e., meningococcus, pneumococcus (eg., N. meningitidis, S. pneumoniae) or H. influenzae.
* Participants with sepsis or active systemic bacterial, viral (including COVID-19) or fungal infection within 14 days prior to study treatment administration.
* Kidney, bone marrow transplant (BMT)/hematopoietic stem cell transplant (HSCT), heart, lung, small bowel, pancreas, liver transplantation or any other cell or solid organ transplantation
* Female patients who are pregnant or breastfeeding, or intending to conceive during the course of the study
* Any medical condition deemed likely to interfere with the patient's participation in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-07-21 (Estimated); Study Completion 2029-07-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants free of TMA manifestation | 12 months
  Absence of thrombotic microangiopathy (TMA) manifestation, without use of anti-C5 antibody, during the 12 months of iptacopan treatment following the switch of treatment from an anti-C5 antibody to iptacopan treatment.

SECONDARY OUTCOMES:
Percentage of participants free of TMA manifestation in study participants with functionally significant mutations in complement genes or positive anti FH antibodies | 12 months, 24 months
  Absence of thrombotic microangiopathy (TMA) manifestation in study participants with functionally significant mutations in complement genes or positive anti FH antibodies, without the use of anti-C5 antibody during iptacopan treatment following the switch of treatment from an anti-C5 antibody to iptacopan treatment.
Percentage of participants free of TMA manifestation | 24 months
  Absence of thrombotic microangiopathy (TMA) manifestation, without use of anti-C5 antibody, during the 24 months of iptacopan treatment following the switch of treatment from an anti-C5 antibody to iptacopan treatment.
Time to TMA manifestation | 12 months, 24 months
  Time to thrombotic microangiopathy (TMA) manifestation
Change from baseline in platelets | Baseline, month 12, month 24
  Change from baseline in platelets at month 12 and month 24.
Change from baseline in LDH | Baseline, month 12, month 24
  Change from baseline in lactate dehydrogenase (LDH) at month 12 and month 24.
Change from baseline in hemoglobin | Baseline, month 12, month 24
  Change from baseline in hemoglobin at month 12 and month 24.
Change from baseline in serum creatinine | Baseline, month 12, month 24
  Change from baseline in serum creatinine at month 12 and month 24.
Change from baseline in UPCR | Baseline, month 12, month 24
  Change from baseline in urine protein to creatinine ratio (UPCR) at month 12 and month 24.
Change from baseline in eGFR | Baseline, month 12, month 24
  Change from baseline in estimated glomerular filtration rate (eGFR) at month 12 and month 24.
Change from baseline in CKD stage | Baseline, month 12, month 24
  Change from baseline in chronic kidney disease (CKD) stage at month 12 and month 24.
Number of participants who require dialysis | month 12 and month 24
  Dialysis requirement status (Yes/ No)
Percentage of participants with TMA related events. | month 12 and month 24
  Percentage of participants with thrombotic microangiopathy (TMA) related events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- China (3):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Kiel
- Italy (3):
  - Novartis Investigative Site, Ranica, BG
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Japan (2):
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
- Spain (5):
  - Novartis Investigative Site, Santiago Compostela, Galicia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Kocaeli, Izmit
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Mersin, Yenisehir
- United Kingdom (3):
  - Novartis Investigative Site, Newcastle upon Tyne, Tyne and Wear
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com